CLINICAL TRIAL: NCT00643916
Title: Safety and Immunogenicity of a Tetravalent (A, C, Y, and W-135) Meningococcal Diphtheria Toxoid Conjugate Vaccine (TetraMenD) In Toddlers 9 to 18 Months of Age
Brief Title: Study of a Tetravalent Meningococcal Diphtheria Toxoid Conjugate Vaccine in Toddlers 9 to 18 Months of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTA26
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Results first posted 2010-01-08 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-01

CONDITIONS: Meningitis; Meningococcal Infection
Keywords: Meningitis; Meningococcal Infection
MeSH Terms: conditions — Meningitis; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Vaccinated at Age 9 and 12 Months (Experimental): Participants received Menactra® vaccine at 9 and 12 Months of age
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Protein Conjugate (Menactra®)
- Vaccinated at Age 9 and 15 Months (Experimental): Participants received Menactra® vaccine at 9 and 15 Months of age
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Protein Conjugate (Menactra®)
- Vaccinated at Age 12 and 15 Months (Experimental): Participants received Menactra® vaccine at Age 12 and 12 Months of age
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Protein Conjugate (Menactra®)
- Vaccinated at Age 15 Months (Experimental): Participants received Menactra® vaccine at 15 Months of age
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Protein Conjugate (Menactra®)
- Vaccinated at Age 18 Months (Experimental): Participants received Menactra® vaccine at 18 Months of age
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Protein Conjugate (Menactra®)
- Vaccinated at Age 3 Years to <6 Years (Active Comparator): Participants received Menomune® vaccine at Age 3 years to <6 years of age
  Interventions: Biological: A/C/Y/W-135, Meningococcal Polysaccharide Vaccine (Menomune®)

INTERVENTIONS:
Biological: Meningococcal Polysaccharide Diphtheria Protein Conjugate (Menactra®) — 0.5 mL, Intramuscular (at age 9 and 12 months)
  Other Names: Menactra®
  Arms: Vaccinated at Age 9 and 12 Months
Biological: Meningococcal Polysaccharide Diphtheria Protein Conjugate (Menactra®) — 0.5 mL, Intramuscular (at age 9 and 15 months)
  Other Names: Menactra®
  Arms: Vaccinated at Age 9 and 15 Months
Biological: Meningococcal Polysaccharide Diphtheria Protein Conjugate (Menactra®) — 0.5 mL, Intramuscular (at age 12 and 15 months)
  Other Names: Menactra®
  Arms: Vaccinated at Age 12 and 15 Months
Biological: Meningococcal Polysaccharide Diphtheria Protein Conjugate (Menactra®) — 0.5 mL, Intramuscular (at age 15 months)
  Other Names: Menactra®
  Arms: Vaccinated at Age 15 Months
Biological: Meningococcal Polysaccharide Diphtheria Protein Conjugate (Menactra®) — 0.5 mL, Intramuscular (at age 18 months)
  Other Names: Menactra®
  Arms: Vaccinated at Age 18 Months
Biological: A/C/Y/W-135, Meningococcal Polysaccharide Vaccine (Menomune®) — 0.5 mL, Subcutaneous (at 3 years to <6 years of age)
  Other Names: Menomune®
  Arms: Vaccinated at Age 3 Years to <6 Years

SUMMARY:
The purpose of this clinical trial is to describe the safety and immunogenicity of one or two doses of Menactra® (TetraMenD) administered in children less than 2 years of age.

Primary Objective:

To describe the immunogenicity profile of one or two doses of Menactra® (TetraMenD) when administered to subjects aged 9, 12, 15, or 18 months in comparison to the immunogenicity of one dose of Menomune® when administered to children aged 3 years to <6 years of age.

DETAILED DESCRIPTION:
This is a Phase II, open-label, parallel, exploratory, multi-center study in healthy toddlers.

ELIGIBILITY:
Inclusion Criteria :

* Aged either 9, 12, 15 or 18 months of age or 3 to < 6 years of age on the day of inclusion.
* Informed consent form that has been approved by the site's Institutional Review Board (IRB) and signed by the parent or legal guardian
* Able to attend all scheduled visits and to comply with all trial procedures

Exclusion Criteria :

* History of a serious chronic disease that could interfere with trial conduct or completion.
* Known or suspected impairment of immunologic function.
* Acute medical illness with or without fever within the last 72 hours, or rectal temperature ≥ 100.4°F (≥ 38.0°C) or axillary temperature ≥ 99.4°F (≥ 37.4°C) on the day of inclusion.
* History of invasive meningococcal disease (confirmed either clinically, serologically or microbiologically) or previous meningococcal vaccination.
* Administration of immune globulin or other blood products within 3 months, or oral or parenteral corticosteroids or other immunosuppressive therapy within the last 6 weeks of the study vaccine. Individuals on a tapering dose schedule of oral steroids lasting < 7 days may be included in the trial as long as they have not received more than one course within the last two weeks prior to enrollment.
* Antibiotic therapy within the 72 hours prior to having any blood sample drawn.
* Received or scheduled to receive any vaccine in the 28-day period prior to receipt of either dose of the study vaccine, or scheduled to receive any vaccination other than influenza vaccination and hyposensitization therapy in the 28-day period after receipt of either dose of the study vaccine. Hyposensitization therapy and influenza vaccination may be received up to two weeks before or after receiving the trial vaccine.
* Suspected or known hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances.
* Thrombocytopenia or a bleeding disorder contraindicating intramuscular vaccination
* Unable to attend one or more of the scheduled visits or to comply with the study procedures.
* Participation in another clinical trial in the 4 weeks preceding enrollment.
* Planned participation in another clinical trial during the present trial period.
* Any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine.

Ages: 9 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 378 (Actual)
Dates: Start 2004-12; Primary Completion 2006-03 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (14):
- United States (14):
  - Little Rock, Arkansas
  - Norwich, Connecticut
  - Atlanta, Georgia
  - Marietta, Georgia
  - Bardstown, Kentucky
  - Baltimore, Maryland
  - Woburn, Massachusetts
  - Akron, Ohio
  - Columbus, Ohio
  - Drexel Hill, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Sellersville, Pennsylvania
  - Kingsport, Tennessee
  - Salt Lake City, Utah

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 10 December 2004 to 14 May 2005 in 15 medical centers in the US
Pre-assignment Details: A total of 378 participants that met the inclusion and exclusion criteria were enrolled, 369 were vaccinated.
Groups:
- Vaccinated at Age 9 and 12 Months: Participants received Menactra vaccine at 9 and 12 months of age
- Vaccinated at Age 9 and 15 Months: Participants received Menactra vaccine at 9 months and 15 months of age
- Vaccinated at Age 12 and 15 Months: Participants received Menactra vaccine at 12 months and 15 months of age
- Vaccinated at Age 15 Months: Participants received Menactra vaccine at 15 months of age
- Vaccinated at Age 18 Months: Participants received Menactra vaccine at 18 months of age
- Vaccinated at Age 3 Years to <6 Years: Participants received Menomune vaccine at age 3 years to <6 years of age
Period: Overall Study
Arm/Group | Vaccinated at Age 9 and 12 Months | Vaccinated at Age 9 and 15 Months | Vaccinated at Age 12 and 15 Months | Vaccinated at Age 15 Months | Vaccinated at Age 18 Months | Vaccinated at Age 3 Years to <6 Years
Started | 55 | 67 | 68 | 62 | 59 | 67
Completed | 51 | 61 | 62 | 60 | 57 | 66
Not Completed | 4 | 6 | 6 | 2 | 2 | 1
Not completed — Protocol Violation | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 2 | 1 | 0 | 1
Not completed — Not Vaccinated | 2 | 2 | 3 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccinated at Age 9 and 12 Months | Vaccinated at Age 9 and 15 Months | Vaccinated at Age 12 and 15 Months | Vaccinated at Age 15 Months | Vaccinated at Age 18 Months | Vaccinated at Age 3 Years to <6 Years | Total
Number analyzed (Participants) | 55 | 67 | 68 | 62 | 59 | 67 | 378
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 55 | 67 | 68 | 62 | 59 | 67 | 378
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 8.9 (0.4) | 8.9 (0.3) | 11.9 (0.3) | 14.9 (0.3) | 17.9 (0.3) | 48.0 (10.3) | 18.7 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 34 | 34 | 23 | 34 | 30 | 179
  Male | 31 | 33 | 34 | 39 | 25 | 37 | 199
Region of Enrollment [Number; unit: participants]
  United States | 55 | 67 | 68 | 62 | 59 | 67 | 378

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥8 Antibody Titers as Measured by Serum Bactericidal Assay Human Complement (SBA-HC) After Each Vaccination.
Time Frame: Day 0 (baseline) and Day 28 post-Vaccinations 1 and 2
Population: Serum Bactericidal Assay Human Complement antibody titers to each of the 4 meningococcal serogroups in the vaccine was evaluated in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vaccinated at Age 9 and 12 Months | Vaccinated at Age 9 and 15 Months | Vaccinated at Age 12 and 15 Months | Vaccinated at Age 15 Months | Vaccinated at Age 18 Months | Vaccinated at Age 3 Years to <6 Years
Number analyzed (Participants) | 40 | 50 | 54 | 55 | 51 | 63
Percentage of Participants
  Meningococcal serogroup A (Baseline) | 38 | 44 | 33 | 40 | 40 | 71
  Meningococcal serogroup A (Post dose 1) | 76 | 67 | 52 | 76 | 65 | 87
  Meningococcal serogroup A (Post dose 2) | 89 | 89 | 85 | 0 | 0 | 0
  Meningococcal serogroup C (Baseline) | 5 | 2 | 0 | 2 | 4 | 8
  Meningococcal serogroup C (Post dose 1) | 83 | 85 | 85 | 86 | 77 | 49
  Meningococcal serogroup C (Post dose 2) | 100 | 100 | 100 | 0 | 0 | 0
  Meningococcal serogroup Y (Baseline) | 3 | 0 | 2 | 2 | 8 | 8
  Meningococcal serogroup Y (Post dose 1) | 21 | 24 | 35 | 33 | 47 | 66
  Meningococcal serogroup Y (Post dose 2) | 95 | 94 | 96 | 0 | 0 | 0
  Meningococcal serogroup W-135 (Baseline) | 3 | 0 | 0 | 2 | 0 | 10
  Meningococcal serogroup W-135 (Post dose 1) | 24 | 27 | 18 | 42 | 36 | 61
  Meningococcal serogroup W-135 (Post dose 2) | 92 | 92 | 96 | 0 | 0 | 0

2. Other Pre Specified Outcome: Percentage of Participants Reporting Solicited Local and Systemic Reactions Within Days 0 to 7 Post-Vaccination.
Description: Solicited local reactions: Redness, Swelling, and Tenderness. Solicited systemic reactions: Fever (temperature), Vomiting, Crying abnormal, Drowsiness, Appetite lost, and Irritability.
Time Frame: Day 0 up to 7 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated study participants, intent-to-treat population.
Measure: Number; unit: Percentage of participants
Arm/Group | Vaccinated at Age 9 and 12 Months | Vaccinated at Age 9 and 15 Months | Vaccinated at Age 12 and 15 Months | Vaccinated at Age 15 Months | Vaccinated at Age 18 Months | Vaccinated at Age 3 Years to <6 Years
Number analyzed (Participants) | 53 | 65 | 65 | 62 | 57 | 67
Percentage of participants
  Any Solicited Injection Site Reaction-Any Dose | 74 | 69 | 65 | 53 | 61 | 55
  Any Solicited Injection Site Reaction - Dose 1 | 62 | 45 | 57 | 53 | 61 | 55
  Grade 3 Solicited Injection Site Reaction - Dose 1 | 0 | 2 | 2 | 0 | 2 | 8
  Any Erythema | 32 | 20 | 34 | 37 | 39 | 33
  Grade 3 Erythema (≥ 2 inches) | 0 | 2 | 2 | 0 | 2 | 2
  Any Swelling | 23 | 8 | 15 | 15 | 23 | 12
  Grade 3 Swelling (≥ 2 inches) | 0 | 0 | 2 | 0 | 2 | 0
  Any Tenderness | 43 | 31 | 37 | 35 | 49 | 48
  Grade 3 Tenderness (cries when inj. limb is moved) | 0 | 0 | 0 | 0 | 0 | 6
  Any Solicited Systemic Reaction-Any Dose | 89 | 84 | 72 | 75 | 72 | 31
  Any Solicited Systemic Reaction Dose 1 | 72 | 75 | 60 | 75 | 72 | 31
  Grade 3 Solicited Systemic Reaction Dose 1 | 9 | 8 | 5 | 12 | 7 | 0
  Any Fever | 23 | 17 | 11 | 18 | 21 | 3
  Grade 3 Fever (≥ 39.6 ºC) | 2 | 3 | 0 | 3 | 0 | 0
  Any Vomiting | 17 | 20 | 11 | 8 | 11 | 5
  Grade 3 Vomiting (≥ 6 episodes per day) | 4 | 0 | 0 | 3 | 0 | 0
  Any Crying Abnormal | 34 | 36 | 28 | 30 | 19 | 13
  Grade 3 Crying Abnormal (> 3 hours) | 4 | 3 | 2 | 2 | 2 | 0
  Any Drowsiness | 40 | 38 | 31 | 35 | 37 | 18
  Grade 3 Drowsiness (difficulty to wake up) | 4 | 0 | 0 | 0 | 4 | 0
  Any Appetite Lost | 28 | 36 | 28 | 37 | 35 | 13
  Grade 3 Appetite Lost (refuses ≥ 3 feeds) | 4 | 2 | 5 | 5 | 0 | 0
  Any Irritability | 60 | 61 | 49 | 57 | 51 | 22
  Grade 3 Irrtability (inconsolable) | 4 | 5 | 3 | 3 | 5 | 0
  Any Solicited Injection Site Reaction - Dose 2 | 63 | 54 | 48 | 0 | 0 | 0
  Grade 3 Solicited Injection Site Reaction - Dose 2 | 2 | 7 | 0 | 0 | 0 | 0
  Any Erythema | 29 | 36 | 23 | 0 | 0 | 0
  Grade 3 Erythema (≥ 2 inches) | 0 | 2 | 0 | 0 | 0 | 0
  Any Swelling | 25 | 20 | 11 | 0 | 0 | 0
  Grade 3 Swelling (≥ 2 inches) | 0 | 3 | 0 | 0 | 0 | 0
  Any Tenderness | 52 | 42 | 37 | 0 | 0 | 0
  Grade 3 Tenderness (cries when inj. limb is moved) | 2 | 3 | 0 | 0 | 0 | 0
  Any Solicited Systemic Reaction Dose 2 | 83 | 56 | 53 | 0 | 0 | 0
  Grade 3 Solicited Systemic Reaction Dose 2 | 13 | 9 | 5 | 0 | 0 | 0
  Any Fever | 28 | 15 | 10 | 0 | 0 | 0
  Grade 3 Fever (≥ 39.6 ºC) | 2 | 0 | 0 | 0 | 0 | 0
  Any Vomiting | 19 | 10 | 8 | 0 | 0 | 0
  Grade 3 Vomiting ≥ 6 episodes per day) | 0 | 2 | 0 | 0 | 0 | 0
  Any Crying Abnormal | 50 | 29 | 27 | 0 | 0 | 0
  Grade 3 Crying Abnormal (> 3 hours) | 6 | 2 | 2 | 0 | 0 | 0
  Any Drowsiness | 42 | 25 | 18 | 0 | 0 | 0
  Grade 3 Drowsiness (difficulty to wake up) | 0 | 2 | 0 | 0 | 0 | 0
  Any Appetite Lost | 31 | 32 | 29 | 0 | 0 | 0
  Grade 3 Appetite Lost (refuses ≥ 3 feeds) | 0 | 3 | 0 | 0 | 0 | 0
  Any Irritability | 63 | 42 | 44 | 0 | 0 | 0
  Grade 3 Irritability (inconsolable) | 10 | 7 | 5 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for 6 months post-vaccination.
Arm/Group | Vaccinated at Age 9 and 12 Months | Vaccinated at Age 9 and 15 Months | Vaccinated at Age 12 and 15 Months | Vaccinated at Age 15 Months | Vaccinated at Age 18 Months | Vaccinated at Age 3 Years to <6 Years
Serious Adverse Events (participants affected / at risk) | 0/53 | 3/65 | 4/65 | 1/61 | 5/57 | 3/67
Other Adverse Events (participants affected / at risk) | 37/53 | 50/65 | 48/65 | 34/61 | 33/57 | 21/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccinated at Age 9 and 12 Months (N=53) | Vaccinated at Age 9 and 15 Months (N=65) | Vaccinated at Age 12 and 15 Months (N=65) | Vaccinated at Age 15 Months (N=61) | Vaccinated at Age 18 Months (N=57) | Vaccinated at Age 3 Years to <6 Years (N=67)
Granulocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia adenoviral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccinated at Age 9 and 12 Months (N=53) | Vaccinated at Age 9 and 15 Months (N=65) | Vaccinated at Age 12 and 15 Months (N=65) | Vaccinated at Age 15 Months (N=61) | Vaccinated at Age 18 Months (N=57) | Vaccinated at Age 3 Years to <6 Years (N=67)
Conjunctivitis (Eye disorders) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 3 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 9 (12) | 13 (18) | 8 (9) | 6 (7) | 8 (9) | 2 (2)
Teething (Gastrointestinal disorders) | 8 (10) | 13 (22) | 17 (23) | 5 (6) | 5 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (5) | 3 (3) | 2 (2) | 3 (3) | 0 (0)
Injection site haemorrhage (General disorders) | 3 (3) | 9 (9) | 7 (9) | 0 (0) | 4 (4) | 7 (7)
Pyrexia (General disorders) | 6 (6) | 13 (16) | 7 (8) | 3 (3) | 7 (7) | 4 (4)
Otitis media (Infections and infestations) | 3 (3) | 13 (15) | 6 (6) | 5 (5) | 4 (4) | 1 (1)
Otitis media acute (Infections and infestations) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 4 (4) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 13 (13) | 8 (9) | 6 (6) | 5 (5) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 12 (14) | 12 (16) | 7 (7) | 7 (7) | 9 (9)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 7 (7) | 5 (8) | 0 (0) | 5 (5) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 6 (6) | 10 (12) | 7 (7) | 2 (2) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6) | 3 (4) | 3 (3) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 4 (4) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications